CLINICAL TRIAL: NCT03833115
Title: A Pilot Descriptive Study On The Spermicidal Efficacy Of A Vaginal Gel Containing Or Not Sodium Lauryl Sulfate In Healthy Women And Their Male Partners
Brief Title: Spermicidal Efficacy Of A Vaginal Gel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Michel G. Bergeron, MD FRCPC, Professor, Laval University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CRI-INV.15
Record Dates: First submitted 2019-01-22; First posted 2019-02-06 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Contraception

STUDY DESIGN:
Intervention Model Description: Pilot descriptive study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- vaginal gel containing sodium lauryl sulfate (Experimental)
  Interventions: Other: vaginal gel containing or not sodium lauryl sulfate

INTERVENTIONS:
Other: vaginal gel containing or not sodium lauryl sulfate — Prevention
  Other Names: Prevention

SUMMARY:
There is an urgent need to develop non-hormonal innovative preventive measures under the control of women that can prevent unintended pregnancy. Based on our experimental data, the use of a gel formulation containing SLS could represent a potent and safe topical vaginal spermicide. The impact of such a preventive tool on public health will be enormous. After successfully completing supportive Phase I/II safety trials, the next step is a prospective pilot clinical trial to evaluate the safety and effectiveness of our gel formulation as a spermicidal agent and for preventing unintended pregnancy in healthy women.

DETAILED DESCRIPTION:
Study objectives (Outcomes):

The primary objective (Primary outcome) of this clinical trial is to evaluate the spermicidal efficacy in vitro and in post-coital test of gel formulation containing or not 2% SLS, when applied once intravaginally in healthy volunteers (women with their stable male sexual partners).

The secondary objective (Secondary outcome) of the study is to evaluate the safety and preliminary efficacy in preventing pregnancy of the gel formulation containing 2% SLS when used repeatedly before each sexual intercourse for a period of 3 months.

Study design: Pilot trial First phase- During volunteers screening for eligibility, male sexual partners will submit sperm samples; half of the sperm sample will be used for spermogram, and the other half of the sperm sample will be used (if normal spermogram) for in vitro testing of the spermicidal efficacy of the gel formulation components. If eligible, the man and his eligible female sex partner will be enrolled. Eligible women of the eligible male sex partners will have one vaginal gel application up to 30 min before planned sexual intercourse (vaginal penile penetration) with male ejaculating inside the vagina. Women will come to the clinic within a maximum of 12h period after the sexual intercourse for post-coital test. The gel must not be applied during menstrual period. The use of other vaginal products and male condom by participants is prohibited during the study period. A diary will be given to participants to record information concerning the internal use, if any, of any vaginal product (including tampons). This pilot trial will be performed in 1 center at the facilities of the Clinical Research of the CHU de Québec-Université Laval, CHUL.

Second phase- Couples agreeing to use the product repeatedly will continue to use the gel-SLS before each and every sexual intercourse, except during menstruation, for a period of 3 months. Women will report safety parameters after each vaginal use of the gel-SLS and will be followed regularly at the facilities of the Clinical Research of the CHU de Québec-Université Laval, CHUL.

ELIGIBILITY:
Inclusion Criteria:

Woman

1. Healthy woman seeking to space or delay pregnancy aged between 18 and 49 years
2. Sexually active
3. Willing to give written informed consent to participate in the trial
4. Normal physical and gynecological examination
5. Negative urine pregnancy test at screening
6. Willing to engage in planned heterosexual vaginal intercourse with ejaculation inside the vagina
7. Female participant in first phase of the study must be already using and agreeing continuous use of a reliable method of contraception defined as use of hormonal contraception (pill, patch or injection, in accordance with the approved product label) during treatment with the study product and must agree to maintain the contraceptive method for at least 2 weeks after discontinuation of study product if not participating in second phase of the study. If the female participant participates in the second phase of the study, she must stop using the method of contraception during product application and use only the test product provided (vaginal gel-SLS).

Man

1. Healthy man aged 18 years and older
2. Sexually active
3. Normal spermogram at inclusion
4. Normal physical examination
5. Willing to give written informed consent to participate in the trial
6. Willing to engage in planned heterosexual vaginal intercourse with ejaculation inside the vagina for post coital test.

Exclusion Criteria:

Woman

1. Abnormal physical/gynecological examination
2. Pregnant at enrolment
3. Lactating or breastfeeding
4. History of vaginitis during the last 3 months
5. History of using vaginal medications during the last 3 months
6. History of STIs (genital herpes, HIV, gonorrhea, chlamydiasis, syphilis, vulvo-vaginal or cervical HPV) during the last 12 months
7. STIs at time of screening
8. Abnormal laboratory findings with clinical significance
9. Allergy to applicator material (polyethylene), to gel polymer (polyoxyethylene-polyoxypropylene)
10. History of toxic shock syndrome (TSS)
11. Use of other contraceptive methods during the study period other than the ones accepted in the study including intrauterine device (IUD), diaphragm, spermicide, contraceptive ring and fertility awareness methods (first phase of the study, no contraception during the second phase)
12. Post-menopausal (12 months of spontaneous amenorrhea and ≥40 years of age) or physically incapable of becoming pregnant with documented permanent sterilization or history of infertility without anterior pregnancy.
13. Women seeking for efficient contraception
14. Current enrolment in any other clinical trial involving investigational drug, vaccine or medical device.
15. Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant or that could prevent, limit, or confound the protocol specified assessments.

Man

1. Abnormal physical examination
2. Abnormal spermogram
3. Surgical sterilization
4. History of urinary infections during the last 3 months
5. History of STIs (genital herpes, HIV, gonorrhea, chlamydiasis, syphilis, HPV) during the last 12 months
6. STIs at time of screening
7. Abnormal laboratory findings with clinical significance
8. Allergy to gel polymer (polyoxyethylene-polyoxypropylene)
9. Current enrolment in any other clinical trial involving investigational drug, vaccine or medical device.
10. Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant or that could prevent, limit, or confound the protocol specified assessments.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — vaginal product for women and their male sexual partners
Enrollment: 30 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2020-12-04 (Actual)

PRIMARY OUTCOMES:
Measuring motility of spermatozoides in vitro in presence of gel or gel-SLS, and in post-coital test after using gel or gel-SLS | 3-6 months
  * First, the motility of spermatozoides (progressive, non-progressive, or non-motile) in vitro in presence of gel, gel-SLS will be measured.
  * Second, the motility of spermatozoides in post-coital test after single intravaginal application of gel or gel-SLS will be measured in women.

SECONDARY OUTCOMES:
Recording pregnancy occurrence after using gel-SLS | 3 months
  Recording pregnancy (no. of pregnant women) after the intravaginal application of the gel-SLS before each sexual intercourse for a period of 3 months.
Recording adverse events (AE) after using gel-SLS | 3 months
  Recording AE (general and genital AE) after the intravaginal application of the gel-SLS before each sexual intercourse for a period of 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Michel Bergeron, Québec, Canada